CLINICAL TRIAL: NCT05828199
Title: Comparative Evaluation The Effect of Intraoperative Infusion of Dexmedetomidine Versus Low Dose Ketamine on Pain and Inflammatory Biomarkers in Patients Undergoing Nasal Surgery
Brief Title: The Effect of Intraoperative Infusion of Dexmedetomidine Versus Low Dose Ketamine
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Hegazy, Resident of Anesthesia, intensive care and pain management Faculty of Medicine - Al-Azhar University, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ahmed Hegazy
Record Dates: First submitted 2023-04-13; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Nasal Polyps; Nasal Septum, Irregular; Functional Endoscopic Sinus Surgery
MeSH Terms: conditions — Nasal Polyps | interventions — Ketamine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedtomidine group (Active Comparator): About 40 patients will receive bolus dose of dexmedetomidine 0.5-1 μg/kg in 100 mL of normal saline over 10 minutes then, continuous infusion dose of dexmedetomidine 0.2 ug/kg/hr.
  Interventions: Drug: Dexmedetomidine
- ketamin group (Active Comparator): About 40 patients will receive a ketamine bolus dose (0.3 mg/kg IV slowly), then continuous infusion dose of ketamine (0.2 mg/kg/hr).
  Interventions: Drug: Ketamine Hydrochloride

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Comparing between dexmedetomidine versus low dose ketamine infusion in patients undergoing nasal and paranasal sinus surgery as regard, intraoperative hemodynamic stability, blood loss, perioperative opioid requirements, Stress response evaluation through the measurement of serum level of cortisol, IL-6, blood glucose and CRP.
  Arms: ketamin group
Drug: Dexmedetomidine — bolus dose of dexmedetomidine 0.5-1 μg/kg in 100 mL of normal saline over 10 minutes then, continuous infusion dose of dexmedetomidine 0.2 ug/kg/hr
  Arms: Dexmedtomidine group

SUMMARY:
Comparing between dexmedetomidine versus low dose ketamine infusion in patients undergoing nasal and paranasal sinus surgery as regard, intraoperative hemodynamic stability, blood loss, perioperative opioid requirements, Stress response evaluation through the measurement of serum level of cortisol, IL-6, blood glucose and CRP.

DETAILED DESCRIPTION:
The primary objective of anesthesia is balancing the patient's hemodynamics with the best possible surgical outcome. In modern anesthesia, a multimodal approach to balanced anesthesia is targeted with combined general anesthetics and systemic drugs.

Trans-nasal endoscopic surgery (TNES) is a helpful diagnostic and therapeutic modality in paranasal sinus diseases. TNES are associated with signiﬁcant intraoperative bleeding, pain, epistaxis, and transient headaches .

Intra-operative surgical site bleeding is one major complication and all anesthetic techniques pursue the objective to reduce it to achieve better precision, reduced operative time, and faster postoperative wound healing.

Topical medications, surgical positioning, nasal packing, inhalational anesthetics, and systemic drugs are some of the documented methods.

Controlled hypotension is one of the methods to control bleeding. It reduces blood loss, enhances the operative ﬁeld quality (dryness) and studies on hypotensive anesthesia have shown a statistically signiﬁcant reduction in blood loss .

Several systemic drugs have been used to achieve controlled hypotension. However, they have their own set of limitations .

Dexmedetomidine, a highly selective α2 adrenoreceptor agonist, has anxiolytic, sedative, anesthetic, and analgesic properties. It has limited side effects in terms of respiratory depression. Because of these favorable properties, it is commonly used in a wide variety of procedures .

Dexmedetomidine is a relatively new drug approved at the end of 1999 by the Food and Drug Administration (FDA) for humans use for short-term sedationand analgesia (<24 hours) in the intensive care unit (ICU). Dexmedetomidine is a useful sedative agent with analgesic properties, hemodynamic stability and ability to recover respiratory function in mechanically ventilated patients facilitating early weaning .

Ketamine hydrochloride, a well-known anesthetic agent, has been in clinical use for more than four decades . Its antinociceptive-hypnotic effects are most likely the result of the noncompetitive antagonism at the N-methyl-D-aspartate (NMDA) receptor of the central nervous system .

Ketamine is used as an analgesic in low doses and as an anesthetic in high doses. It is suggested that ketamine maintains analgesia and reduces postoperative opioid use, whether used alone or in combination with other anesthetic agents, The perioperative use of ketamine in surgery with moderate-to-severe postoperative pain is recommended by the American Society of Regional Anesthesia and Pain Medicine, American Academy of Pain Medicine, and American Society of Anesthesiologists.

Cytokines regulate the host response to infection, the immune response, inflammation, and trauma. Surgical stress has been reported to be associated with elevated cytokines response. IL-6 is highly expressed during inflammatory responses to conditions of stress, and can be used to assess the severity of surgical trauma.

The stress response to surgery is characterized by increased secretion of pituitary hormones and activation of the sympathetic nervous system, For example, release of corticotrophin from the pituitary stimulates cortisol secretion from the adrenal cortex .

ELIGIBILITY:
Inclusion Criteria:

* • Between 21 and 40 years of age, they with American Society of Anesthesiologists (ASA) physical status I-II and undergoing nasal and paranasal sinus surgery.

Exclusion Criteria:

* • Refusal to join the study.

  * Allergy to the drugs used in the study.
  * Drug and/or alcohol abuse.
  * Mental and psychiatric disorders.
  * Emergency operations.
  * Patients with systemic illnesses (eg, hypertension [ SBP >160 mm Hg], diabetes mellitus.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
The postoperative pain | from 0 hours to 24 hours after the procedure
  Assessed by VAS score.As (VAS:0-10, where 0 = no pain, and 10 = worst possible pain). Before surgery, all patients will be a short education about VAS.

CONTACTS AND LOCATIONS:
Overall Officials: Essam Ali, Professor, Study Chair — Al-Azhar University, Faculty of medicine for boys
Locations (1):
- Faculty of Medicine, Al-Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided